CLINICAL TRIAL: NCT03295799
Title: Patient-Centred Care for Warfarin Management: A Pilot Study to Transition Care to High Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052090
Record Dates: First submitted 2017-09-18; First posted 2017-09-28 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Self-Management (Experimental): Patients will go through a preparatory phase (creation of warfarin dosing chart, process for documentation and retrieval of labs), a practical training phase (formulate warfarin management plan with support) and then perform patient-self management of their own warfarin.
  Interventions: Other: Patient Self-Management
- Anticoagulation Clinic Care (No Intervention): Patients will not have their care altered, and will continue to be managed by our Anticoagulation Clinic.

INTERVENTIONS:
Other: Patient Self-Management — Patient will manage their own warfarin therapy.
  Arms: Patient Self-Management

SUMMARY:
Warfarin remains the only oral anticoagulant effective in preventing stroke and valve thrombi for patients having mechanical heart valves (MHVs). Within Edmonton, Alberta, our pharmacist-directed and staffed Anticoagulation Clinic (AC) is referred all MHVs implanted, and now has ~450 active patients. The AC mandate is to work with patients to ensure they have a thorough understanding of their warfarin therapy and the factors that may impact its control. In European countries patients are often taught to manage their own warfarin therapy (=Patient Self-Management [PSM]) and achieve good warfarin control and outcomes. Despite advocating for a patient-centred approach for healthcare delivery in Alberta, no established programs (or funding models) exist to teach and provide ongoing support for PSM in North America. The patient population (namely MHVs) served at our AC offers a unique opportunity to implement PSM given they are already aware of their therapy and only require some extra training and support to assume their own management. While it is anticipated that an increase in pharmacist AC resources would be necessary to teach patients to self-manage, the establishment of a PSM program has the potential to free up AC resources in the long-term, allowing more patients to be managed with reducing waiting times for the AC. With infrastructure in place, the AC could serve as a centre of excellence for PSM, accepting referrals for this level of care from across the province. Given the patient-centred approach to care delivery in Alberta, it remains prudent to assess patient acceptability to the PSM approach to anticoagulation care delivery. As such, the primary objective of this randomized pilot study is to assess the effect of PSM compared to AC care on quality of life. Our results will inform a larger scale future trial.

DETAILED DESCRIPTION:
50 patients will receive a cover letter outlining their random selection for this study, along with the patient information sheet and consent form (with a return addressed, postage paid envelope). Patients will be encouraged to contact the AC and speak with the Principal Investigator (TB) regarding the research study, and all questions will be addressed. We will continue this mailing process until a total of 50 patients have consented to study. PSM within the context of this study may use either POC technology or standard venipuncture with the patient accessing the laboratory for results. After receipt of consent, patients will be required to pass a foundational exam (outlining the basics of anticoagulation therapy, most of which should be simple review for the patients managed within our AC).4,10 Upon successfully passing this multiple choice exam, patients will be randomized to AC care (with no changes implemented) or to PSM.

PSM Phase I: Preparatory Phase of Patient Training (~6weeks) During the initial preparatory phase lasting 6 weeks + 2 weeks, the AC will create a patient specific warfarin dosing nomogram, discuss the same with the patient and ensure clear understanding, while working through various scenarios with the patient (Appendix 1). The AC will ensure the patient has an established system to both retrieve INR results (via POC technology or standard venipuncture) as well as to document the INR results, warfarin dosing, any pertinent assessment factors, and next date to test the INR. The AC will empower the patient to be proactive with coming up with warfarin dose changes during this preparatory phase.

PSM Phase II: Patient Practical Training:

The AC will enrol the patient into the PSM practical training phase (lasting 3 months + 1 month). At this time, the patient will retrieve their result and establish a future warfarin dose and follow-up plan. This information will be transmitted to a single AC team member. Contact with anotherdiscussed with an AC team member and the ultimate dosing decision will be tracked to ascertain concordance of the patient's original plan to what was implemented during the follow-up visit with the to perform standard AC teamcare and management will occur, thereby enabling comparison of the patient's plan and the AC plan. During this phase, the AC plan will be implemented. At the end of this phase, patients must pass a multiple choice exam that provides practical cases targeting warfarin dose adjustment with next scheduled follow-up visit, and will then be positioned into the PSM arm of the study.

Patient Self-Management During the PSM phase (6 months +/- 1 month), contact will occur with the AC monthly to retrieve INR results and warfarin dose adjustments (information from the patient-based charting system). Key points of contact between the patient and the AC will be required, such as: INR results either > 5.0 or 0.5 INR units below the lower limit of their desired target INR range, initiation of interacting medications, illness, etc. Patients not demonstrating the ability to self-manage their own warfarin therapy will be encouraged to cross-over to AC care. At the end of 6 months, patient choice of AC care or PSM will be identified.

ELIGIBILITY:
Inclusion Criteria:

* mechanical heart valve as the indication for warfarin
* > 16 years of age
* Warfarin therapy managed by the AC for at least the preceding 6 months
* Anticipated duration of warfarin therapy to be lifelong
* Previously adherent with medication
* Competence judged by demonstrated ability to use drug-adjustment nomograms

Exclusion Criteria:

* • Severe psychiatric disease

  * Significant language barrier
  * Clinician's judgment that the patient would be a poor candidate for study (with reason specified)
  * Known or anticipated procedure/surgery/intervention in the next year
  * Active participation in another study
  * Lack of access to the internet / email

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
The change in quality of life score (using the validated instruments DASS and Sawicki scale) between PSM and AC care. | 6 months
  Duke Anticoagulation Satisfaction Scale (DASS) and Sawicki Scale

SECONDARY OUTCOMES:
The proportion of patients completing PSM | 9 months
  Beginning from consent and capturing stage at which patients withdrew (if applicable) namely the preparatory and practical training phases or PSM as well as those electing to continue PSM after study
Difference in the time in therapeutic INR range between those randomized to AC care versus PSM. | 6 months
  Time in range will be calculated using the Rosendaal method.
The rate of ER and hospitalization for anticoagulant and non-anticoagulant reasons between AC care and PSM. | 6 months
  presentations to hospital
The amount of time spent by the AC team for the AC group relative to the PSM group. | 9 months
  the number of minutes taken for each arm, as a measure of resource use within the AC team.
Amongst the PSM group, to determine if strategies for self-managing warfarin therapy have made patients do so for other chronic diseases. | 6 months
  a descriptive measure of translation of proactive management
Number of participants in AC care vs PSM that are dead at 5 years. | 5 years following study completion
  mortality measure
Number of encounters in the PSM group that put forward warfarin dosing that is concordant with that of the AC and to provide descriptions of warfarin dose changes. | 3 months
  assessed prior to entering the PSM phase

CONTACTS AND LOCATIONS:
Overall Officials: Tammy Bungard, BSP, PharmD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No